CLINICAL TRIAL: NCT05055492
Title: The School SPIT Study (Saliva to Promote Improved Testing): A Prospective Evaluation of a Home Saliva Testing Program Implemented With a Stepped-wedge Cluster Randomized Design in Elementary Schools in High SARS-CoV-2 Incidence Regions
Brief Title: The School SPIT Study - Elementary Schools in High COVID-19 Incidence Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Principle Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000078377-2
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV2 Infection
Keywords: School Testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a prospective evaluation of a program that is being implemented using a stepped-wedge, cluster randomized design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control period (No Intervention): Schools will start in the control phase (SARS-CoV-2 diagnostic testing at an assessment center, primary care office or acute care center) and transition to the intervention phase at a randomly assigned time point over the course of the study.
- Intervention phase (Active Comparator): Schools will have take home saliva kits available at the school to support SARS-CoV-2 diagnostic testing. Schools will transition to the intervention phase at a randomly assigned time (wedge) over a 6-week period with all schools receiving the program by the end of the study.
  Interventions: Diagnostic Test: Take home saliva kits

INTERVENTIONS:
Diagnostic Test: Take home saliva kits — Saliva kits will be made available at schools for pick up to support symptomatic testing using PCR for students, staff and family members.
  Arms: Intervention phase

SUMMARY:
This study will conduct an evaluation of a program that is being implemented SickKids / Toronto Public Health that provides take-home saliva testing kits in schools. Operationally, there is a planned randomization so that all schools have an equitable chance to receive the intervention at various time periods during the planned operational roll-out, which will require a staggered implementation consistent with the stepped-wedge study design. This study will leverage this chance implementation to do a robust evaluation of the public health intervention. Schools that are not being rolled out to week one, will begin in the "control phase" (testing at an assessment center, primary care or acute care center) and transition to the program "intervention phase" (take home saliva kits available at schools) at a randomly assigned time (wedge) over a 6-week period with all schools receiving the program by the end of the study. The investigators will evaluate the impact of the program on SARS-CoV-2 case identification in schools.

DETAILED DESCRIPTION:
This is a prospective evaluation of a program that is being implemented using a stepped-wedge, cluster randomized design.

Eligible elementary public schools high SARS-CoV-2 incidence regions (quintiles 4 and 5) in Toronto will be randomized. The study will occur over a 7-week period with a minimum of one-week of baseline data (control phase - testing at an assessment center, primary care or acute care center) and then schools will start the program in a stepwise manner (20 crossovers per week) with take-home saliva being available to all 120 schools by the end of the study period. The primary objective of the study is to assess whether the availability of take home saliva kits at schools for symptomatic testing leads to increased diagnosis of SARS-CoV-2 cases in the school.

ELIGIBILITY:
Elementary schools will be included in the evaluation if they are:

* Considered an elementary school by the school board
* Open for in-person learning during the study period
* They have at least 200 students
* Offer at least 4 grades

Exclusion Criteria:

Schools that are middle schools only, that are not open for in-person learning, have fewer than 200 students or are not a complete elementary school (i.e. schools offering independent courses, prep schools with 1-2 grades, elementary schools with < 4 grades) will be excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 Case identification | Weekly measurement over 7 week study period
  The number of cases positive for SARS-CoV-2 in a cohort per week per school

SECONDARY OUTCOMES:
Uptake of take-home saliva kits for testing | Weekly measurement over 7 week study period
  Frequency of use of take-home saliva kits per week per school
Impact on timing of test for symptomatic individuals | Over study 7 week study period
  To assess whether availability of take-home saliva kits at schools leads to earlier testing as measured by duration of symptoms before testing of the symptomatic case
Impact on Secondary Transmission | Over 7 week study period
  To assess whether the availability of take-home saliva kits at schools leads to reduced transmission within exposed cohorts as measured by number of secondary cases identified in exposed cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided